CLINICAL TRIAL: NCT05007301
Title: Geko™ Cross Therapy Registry - Wound An Observational Study for the Post Market Clinical Follow-up of Safety and Patient Outcomes for Patients Undergoing Peroneal Nerve Stimulation by Geko™
Brief Title: Geko™ Cross Therapy Registry - Wound
Acronym: CTR-Wound
Status: Active, not recruiting | Type: Observational
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: FSK-REG-002
Record Dates: First submitted 2021-08-05; First posted 2021-08-16 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Wound; Venous Leg Ulcer; Diabetic Foot Ulcer; Arterial Leg Ulcer
Keywords: geko; wound therapy; medical device; registry
MeSH Terms: conditions — Wounds and Injuries; Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Standard of care: Patients who are receiving the geko device as part of standard of care for wound management
  Interventions: Device: geko device

INTERVENTIONS:
Device: geko device — Neuromuscular electrostimulation of the peroneal nerve, 12h per day, for up to 12 weeks.

SUMMARY:
The geko™ Cross Therapy REGISTRY - Wound is a prospective, observational, anonymised data collection Registry with no experimental treatment that will fulfil an unmet need for an observational Registry to provide long-term clinical data to demonstrate patient benefit and regulatory compliance.

DETAILED DESCRIPTION:
The geko™ Cross Therapy REGISTRY - Wound represents a long-term project to integrate prospectively and systematically collected clinical data on all geko™ W wound devices (or W device variants) used in SC pathways for wound management allowing for the monitoring of patient outcomes during a follow-up period of up to four follow-up visits.

The clinical database collected for the geko™ CTR - Wound will form part of the overall post-market clinical follow-up strategy for the device and post market surveillance to support device safety and performance. There will be up to 50 contributing centres globally. Participants are asked at the time of signing up for the geko™ Cross Therapy REGISTRY - Wound (at the recruitment / baseline visit) to attend as many follow up visits as possible (up to a maximum of 4).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Intact healthy skin at the site of geko™ device application.
3. Willing and able to give written informed consent
4. Presence of an ulcerative wound to the lower leg
5. Identified to receive geko™ therapy as part of their standard care for wound management.

Exclusion Criteria:

1. Pregnancy or breast feeding.
2. Use of any other neuro-modulation device.
3. Current use of TENS in the pelvic region, back or legs
4. Trauma to the lower limbs that would prevent geko™ from stimulating the common peroneal nerve.
5. No response to geko™ therapy i.e., no involuntary rhythmic upward and outward movement of the foot (dorsiflexion) at the maximum tolerable device setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have been identified to receive geko™ therapy as part of their standard care for wound management. All participants must be at least 18 years of age and must be able to provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events | Up to 12 months from study entry
  Obtain frequency of adverse events (AEs) whether device related or not and compare rate to historic and published data i.e., geko™ therapy vs standard care without geko™ therapy
Frequency of serious adverse events | Up to 12 months from study entry
  Obtain frequency of serious AEs (SAEs) whether device related or not and compare rate to historic and published data i.e., geko™ therapy vs standard care without geko™ therapy
Frequency of device deficiencies | Up to 12 months from study entry
  Obtain frequency of Device Deficiencies (DD) and compare rate to historic and published data i.e., geko™ therapy vs standard care without geko™ therapy

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Collarte, Principal Investigator — Central London Community Health Care NHS Trust
Locations (3):
- Northwell Health System, New York, New York, United States
- United Kingdom (2):
  - Central London Community Health Care NHS Trust, London
  - Norfolk Community Health and Care NHS Trust, Norwich

IPD SHARING:
Plan to Share IPD: No